CLINICAL TRIAL: NCT07376213
Title: Investigation of the Effects of Home-Based Exercise Program Applied During Radiotherapy on Posture, Range of Motion, Muscle Strength, Fibrosis, Lymphedema and Swallowing Functions in Patients Diagnosed With Head and Neck Cancer
Brief Title: Effects of a Home-Based Exercise Program During Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Burak Ertürk (Other)
Responsible Party: Sponsor-Investigator, Burak Ertürk, Research Assistant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E-77082166-302.08.01-805534
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer
Keywords: head and neck neoplasms; Radiotherapy; Exercise; Physiotherapy; Lymphedema
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity; Lymphedema

STUDY DESIGN:
Masking Description: This was an open-label study. Outcome assessments and interventions were performed by the same researcher. Statistical analysis was conducted by an independent biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Home-Based Physiotherapy Program (Experimental): Participants in the intervention group will receive instruction in a structured home-based exercise program to be implemented throughout the radiotherapy period. Adherence, technique, and progression will be monitored and reinforced through weekly in-person sessions with a qualified professional.
  Interventions: Procedure: Home-based exercise
- Usual Care / Standard Follow-Up (No Intervention): Participants in the control group will receive only radiotherapy and will not undergo any physiotherapy interventions during this period. At the end of the radiotherapy, both groups will be re-evaluated, and participants in the control group will then be provided with appropriate treatment and home-based exercise programs.

INTERVENTIONS:
Procedure: Home-based exercise — The home-based rehabilitation approach was conducted for the patients, consisting of neck and upper extremity mobilization, strengthening, stretching, and breathing exercises, 5 days a week.
  Arms: Structured Home-Based Physiotherapy Program

SUMMARY:
The purpose of this study is to examine the effects of exercise on individuals with head and neck cancer who are receiving postoperative radiotherapy.

The study is based on three primary hypotheses:

1. Exercise may help reduce or prevent the loss of normal range of motion that can occur during radiotherapy.
2. Exercise may help maintain muscle strength or lead to improvements in muscle strength.
3. Exercise may help maintain or improve postural alignment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of squamous cell carcinoma of the head and neck.
* Undergoing unilateral neck dissection surgery.
* Scheduled to receive curative radiotherapy.
* Age 18 years or older.
* Willingness to participate and ability to comprehend exercise instructions.

Exclusion Criteria:

* Presence of distant metastasis.
* Presence of a tracheostomy.
* History of previous trauma or surgery involving the shoulder or cervical region.
* Neurological disorders affecting upper quadrant function. Recurrence of disease during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Range of Motion | Baseline and Day 25 (end of radiotherapy)
  Range of motion of the cervical region will be assessed using a cervical range of motion (CROM) device, and shoulder range of motion will be assessed using a goniometer, including flexion, extension, lateral flexion, rotation, abduction, and external rotation.

SECONDARY OUTCOMES:
Muscle Strength | Baseline and Day 25 (end of radiotherapy)
  Muscle strength of the cervical and shoulder girdle muscles will be evaluated using manual muscle testing.
Postural Alignment | Baseline and Day 25 (end of radiotherapy)
  Postural alignment will be assessed through observational postural analysis focusing on head, neck, and shoulder alignment.
Fibrosis Severity | Day 25 (end of radiotherapy)
  Radiation-induced fibrosis will be evaluated using a standardized clinical fibrosis grading scale.
Lymphedema | Day 25 (end of radiotherapy)
  Head and neck lymphedema will be assessed using circumferential measurements and/or clinical lymphedema grading.
Swallowing Function | Baseline and Day 25 (end of radiotherapy)
  Swallowing function will be evaluated using a validated swallowing assessment scale (Swal-QoL).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Faculty of Health Sciences, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No